CLINICAL TRIAL: NCT00700544
Title: Adjonction of Androgenotheapy for Post-Remission Treatment of Elderly Patients With Acute Myeloid Leukemia - Results of the Multicenter Goelams SA-2002 Trial.
Brief Title: Treatment Outcome in Elderly Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: French Innovative Leukemia Organisation (Other); BGMT (Unknown)
Responsible Party: CHU Grenoble Pr Jean Jacques SOTTO, GOELAMS BGMT
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LAM SA 2002
Record Dates: First submitted 2008-06-13; First posted 2008-06-18 (Estimated); Last update posted 2008-06-18 (Estimated); Status verified 2008-06

CONDITIONS: AML; Elderly Patients
Keywords: AML; elderly patients; Treatment outcome
MeSH Terms: interventions — Norethandrolone; Induction Chemotherapy; Maintenance Chemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- B (Active Comparator): * Induction therapy Idarubicin, 8mg/m2 d1-5; Cytarabine, 100mg/m2 d1-7 and Lomustine, 200mg/m d1) If CR ou PR
  * maintenance therapy every 3 months = 6 courses of reinduction with :
    -idarubicin (8mg/m2 d1),cytarabine (100mg/m2d1-5 ), subcutaneously
  * between the courses, a continuous regimen of methotrexate and 6-mercaptopurine.
  Interventions: Drug: chemotherapy treatment (see arms)
- A (Experimental): * Induction therapy Idarubicin, 8mg/m2 d1-5; Cytarabine, 100mg/m2 d1-7 and Lomustine, 200mg/m d1) If CR ou PR
  * maintenance therapy every 3 months = 6 courses of reinduction with :
    * idarubicin (8mg/m2 d1),cytarabine (100mg/m2d1-5, subcutaneously)
    * 10 to 20 mg (according to body weigh) of norethandrolone daily
  * between the courses, a continuous regimen of methotrexate and 6-mercaptopurine.
  Interventions: Drug: chemotherapy treatment (see arm) + norethandrolone

INTERVENTIONS:
Drug: chemotherapy treatment (see arm) + norethandrolone — oral form
  Dosage:
  10 mg in patients with a weight < 60 kgs 20 mg in patients with a weight > 60 kgs frequency: every day Duration: 2 years
  Other Names: norethandrolone = nilevar®
  Arms: A
Drug: chemotherapy treatment (see arms) — Induction chemotherapy + maintenance chemotherapy
  Other Names: Induction chemotherapy + maintenance chemotherapy
  Arms: B

SUMMARY:
A multicenter randomized trial evaluating the possible benefit of androgens during post remission therapy in an attempt to improve the outcome of AML in older patients.All patients received the ICL regimen as induction and were randomized to receive, after achieving CR or PR, a maintenance therapy including or not androgens. Patients randomized with androgens additionally received 10 to 20 mg according to body weigh of norethandrolone daily for up to 2 years

DETAILED DESCRIPTION:
* Induction Therapy:

  * Idarubicin, 8mg/m2 d1-5; Cytarabine, 100mg/m2 d1-7 and Lomustine, 200mg/m d1
  * if CR or PR: randomisation = maintenance therapy including or not androgens
* Maintenance therapy :

  * 6 courses of reinduction with idarubicin (8mg/m2 d1) and cytarabine (100mg/m2d1-5, subcutaneously) every 3 months, and, between these courses, a continuous regimen of methotrexate and 6-mercaptopurine.
  * Patients randomized with androgens additionally received 10 to 20 mg according to body weigh of norethandrolone daily for up to 2 years

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 60 years or more
* "de novo" AML according to FAB criteria
* AML with 20% or more myeloid marrow blasts
* signed and dated informed consent
* OMS score < 3
* Life expectancy > 1 month

Exclusion Criteria:

* Patients aged < 60 years
* or AML M3
* or not classificated according to FAB criteria
* or extramedular localisation of AML
* OMS score ≥ 3
* clinical Abnormal Cardiac fonction or with left ejection fraction < 40 %
* abnormal renal function with creatinine clearance < 50/ml/mn/m²
* abnormal hepatic function
* previous cerebral stroke
* previous malignancy : prostate, breast cancer (males)
* PSA dosage > 4
* Any coexisting medical or psychological condition that would pleclude participation in the required study procedures

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2002-06; Primary Completion 2005-04 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study was to assess the ability of androgens to increase DFS. | 3 years

SECONDARY OUTCOMES:
The secondary objective was to improved EFS and OS and to assess side effects and toxicity of androgenotherapy | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jean jacques SOTTO, MD, Principal Investigator — GOELAMS/BGMT; Arnaud PIGNEUX, MS, Principal Investigator — GOELAMS/BGMT; Francis WITZ, MS, Principal Investigator — French Innovative Leukemia Organisation
Locations (1):
- Arnaud PIGNEUX, Pessac, France

REFERENCES:
- [Derived] Pigneux A, Bene MC, Guardiola P, Recher C, Hamel JF, Sauvezie M, Harousseau JL, Tournilhac O, Witz F, Berthou C, Escoffre-Barbe M, Guyotat D, Fegueux N, Himberlin C, Hunault M, Delain M, Lioure B, Jourdan E, Bauduer F, Dreyfus F, Cahn JY, Sotto JJ, Ifrah N. Addition of Androgens Improves Survival in Elderly Patients With Acute Myeloid Leukemia: A GOELAMS Study. J Clin Oncol. 2017 Feb;35(4):387-393. doi: 10.1200/JCO.2016.67.6213. Epub 2016 Oct 24. PMID 28129526